CLINICAL TRIAL: NCT03388580
Title: Predictors for Bronchoalveolar Lavage Recovery Rate Derived From Quantified Computed Tomography
Brief Title: Predictors for Bronchoalveolar Lavage (BAL) Recovery Rate Derived From Quantified Computed Tomography (qCT)
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Frederik Trinkmann, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: qCT - BAL
Record Dates: First submitted 2017-12-24; First posted 2018-01-03 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Interstitial Lung Disease; Pneumonia; Malignant Neoplasm
MeSH Terms: conditions — Lung Diseases, Interstitial; Pneumonia; Neoplasms | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAL: patients undergoing elective bronchoalveolar lavage
  Interventions: Procedure: bronchoalveolar lavage (BAL)

INTERVENTIONS:
Procedure: bronchoalveolar lavage (BAL) — clinically indicated, elective BAL

SUMMARY:
Bronchoalveolar lavage (BAL) is an important diagnostic method. The percentage of fluid extracted after instillation (recovery rate) is crucial for following diagnostic tests. The investigators aimed to compare novel quantified airway parameters from pre-interventional lung computed tomography (CT) with recovery rates to find possible predictive markers.

ELIGIBILITY:
Inclusion Criteria:

* retrospective analysis of all patients undergoing BAL and complete documentation

Exclusion Criteria:

* incomplete documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective BAL with clinical indication.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
recovery rate | 30 minutes
  volume of recovered volume

IPD SHARING:
Plan to Share IPD: No